CLINICAL TRIAL: NCT05850078
Title: Vaginal Microbiome Transplant in Asymptomatic Healthy Volunteers, Who Have Undergone Vaginal Microbiome Screening - a Randomised, Double-blind, Placebo-controlled Three-arm Study
Brief Title: FB101 Intervention in Women Screened to Have Vaginal Dysbiosis (Dyscover-3)
Acronym: Dyscover-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freya Biosciences ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Dyscover-3
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Vaginal Flora Imbalance

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, parallel, 3-arm, placebo-controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, clinical investigators as well as outcome assessors (laboratories) will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FB101 (Experimental): Microbial intervention using product FB101
  Interventions: Other: FB101
- FB101 diluted (Experimental): Microbial intervention using diluted FB101
  Interventions: Other: FB101
- Placebo (Placebo Comparator): Saline water
  Interventions: Other: FB101

INTERVENTIONS:
Other: FB101 — Intervention will test effects on changes to the vaginal microbiome of FB101 versus diluted FB101 versus placebo

SUMMARY:
This study will explore and map the potential shifts in vaginal microbiomes as a consequence of a microbial intervention with product FB101 in healthy, asymptomatic volunteer women screened to have vaginal dysbiosis based on criteria defined by quantitative polymerase chain reaction (qPCR) analysis of a vaginal swab sample.

DETAILED DESCRIPTION:
This study will explore and map the potential shifts in vaginal microbiomes as a consequence of a microbial intervention with product FB101 in healthy, asymptomatic volunteer women screened to have vaginal dysbiosis based on criteria defined by qPCR analysis of a vaginal swab sample. A dose of FB101 will be given on 2 different days and subjects will be followed for changes in their vaginal microbiomes until approximately 3 months after the first FB101 dose. Two different dilutions will be tested of FB101 in 2 different active arms. The study will also have a third arm receiving placebo product. In addition, an antiseptic vaginal wash will be performed before the first dose of FB101/placebo in all 3 study arms. Randomisation ratios will be 1:1:1.

The study includes a screening visit where all criteria for participation are checked and a vaginal swab is obtained to check if pre-defined dysbiosis criteria are met based on qPCR analysis of key vaginal bacterial species. If, and when, all criteria are confirmed, a baseline visit is scheduled to be performed around day 14 in the same menstrual cycle of each individual subject. Besides baseline assessments, the subject is randomised to active FB101 or placebo in a ratio of 1(active, FB101):1(active, diluted FB101): 1(placebo) and the first dose is given. At visit 3 (performed the day after baseline visit the following dose is given.

In total, 5 follow-up visits are scheduled to occur for a period of up to 3 months after the first dose. All follow-up visits will be scheduled to occur around day 14 in the subject's menstrual cycle with one menstrual cycle in between visits. At follow up visits, close safety monitoring will be performed as well as metagenomic sequencing assessment of the microbiota in a vaginal swab.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to give written informed consent.
* Age between ≥18 to ≤45.
* Be generally healthy, as determined by the investigator.
* Be a pre-menopausal woman.
* Meet the following definition of vaginal dysbiosis: combined copy number of Lactobacillus species crispatus, gasseri, and jensenii measured by qPCR, corresponding to less than 10% total relative abundance of Lactobacillus species crispatus, gasseri, and jensenii as measured by metagenomic sequencing.
* Have regular, predictable menstrual cycles of known length or have been amenorrhoeic for at least 3 months due to use of a long-acting progestin or hormonal contraceptives.
* Be willing to be asked questions about personal medical, sexual, and behavioural history.
* Be willing to undergo two vaginal microbiome transplant procedures.
* Be willing to self-collect cervicovaginal secretions and vaginal swab samples.
* Be willing to use one of the following effective methods of contraception throughout the clinical study:

  * Complete abstinence from vaginal intercourse.
  * Have a male sexual partner who is surgically sterilised prior to the screening visit and is the only male sexual partner for that participant.
  * Mechanical barrier (condom or diaphragm), or hormone contraception (contraceptive pill, injections, implant or patch).
* Be willing to completely abstain from vaginal intercourse and receptive oral sex during the eight days from visit 4 (first FB101 dose) to visit 6 (first follow-up).
* Be willing to abstain from vaginal intercourse, unless using condoms free from adjunctive spermicide or lubricant (with a male partner) or dental dams (with a female partner), and receptive oral sex, unless using dental dams, in the time period between visit 3 and visit 8.
* Be willing to avoid taking baths, swimming, or sitting in a hot tub in the time period between visit 3 and visit 8.
* Be willing to abstain from using insertive vaginal feminine products (i.e., tampons, menstrual cups), vaginal cleansing products, spermicides, lubricants, or other vaginal products not approved by the study investigators, and any penetration using fingers or sex toys into the vagina, in the time period between visit 3 and visit 8.

Exclusion Criteria:

* Participants who are post-menopausal, defined as more than 12 consecutive months of amenorrhea without another known cause than use of long-acting progestin or hormonal contraceptives.
* Participants who are pregnant, breastfeeding and/or have been pregnant within the last two months.
* Users of any hormonal or non-hormonal intrauterine device (IUD).
* Participants who have HIV/AIDS or other immunodeficiency.
* Participants who test positive at screening for HIV, chlamydia, gonorrhoea, Mycoplasma genitalium, and/or Trichomonas vaginalis. Potential participants may be re-screened if they receive successful treatment at their own medical provider.
* Participants who have received treatment involving experimental drugs less than 30 days prior to this study.
* Participants who have undergone some sort of procedure involving trauma to the cervix within the last month prior to screening (i.e., IUD removal, cervical cryotherapy, or cervical laser treatment).
* Participants with any known condition requiring regular use of antibiotics, that would suggest the participant is likely to require antibiotic treatment during the study.
* Systemic and/or vaginally applied antibiotic use within the last month prior to screening.
* Participants with new (<3 months) use of long-acting hormonal treatments. Participant may be enrolled if stable (>3 months) or existing therapy as determined by the investigator.
* Participants with any social, medical, or psychiatric condition that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
* Participants with a history of drug or alcohol abuse that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
* Participants with a history of gynaecological cancers, gynaecological conditions, or surgical gynaecological medical history, which, in the opinion of the investigator, precludes participation.
* Participants with abnormal finding on screening examination, which, in the opinion of the investigator, precludes participation.
* Participants with clinically relevant abnormalities in the cervix or uterine cavity that could interfere with the collection of endometrial fluid.
* Participants with history of hypersensitivity/allergic reactions to the antiseptic active component or its ingredients.
* Participants who have previously received FB101 as part of a clinical study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 97 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Changes in relative abundance of vaginal lactobacilli species | from baseline to 2 months after first dose
  The change in vaginal microbiome of the active arm participants (FB101 and diluted FB101) versus placebo participants in terms of the combined relative abundance of the vaginal Lactobacillus species crispatus, gasseri and jensenii measured by metagenomic sequencing of vaginal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus McCarthy, PhD, MD, Principal Investigator — Atlantia Clinical Trials
Locations (1):
- Atlantia Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No